CLINICAL TRIAL: NCT00650507
Title: Clinical and Genomic Responses to Open Heart Surgery: A Randomized Controlled Trial of the Effects of Remote Ischemic Preconditioning
Brief Title: Clinical and Genomic Responses to Open Heart Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian McCrindle, Staff Cardiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 1000011898
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Ischemia-reperfusion (IR) Injury
Keywords: children; cardiac surgery; remote ischemic preconditioning; SHAM; ischemia-reperfusion
MeSH Terms: conditions — Wounds and Injuries | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)
- 2 (Active Comparator)
  Interventions: Procedure: SHAM

INTERVENTIONS:
Procedure: Remote ischemic preconditioning (RIPC) — The RIPC stimulus will be delivered in the OR prep room after the induction of anesthesia (while the anesthesiologist and staff are inserting vascular cannulae and preparing the patient for surgery). Whenever possible, the left lower limb will be selected for delivery of the stimulus. An appropriate sized cuff will be selected and connected to a hand aneroid sphygmomanometer. A second cuff and hand aneroid sphygmomanometer will be placed beside the one connected to the study subject. The cuff on the limb will be inflated and deflated to provide a total of four cycles of limb ischemia and reperfusion.
  Arms: 1
Procedure: SHAM — For this group, the procedure will be identical for that described for the RIPC stimulus, with the exception that the blood pressure cuff placed on the subject will not be inflated, but the second cuff, that has been placed beside, will be inflated.
  Arms: 2

SUMMARY:
This study will be the first large scale randomized study of remote ischemic preconditioning (RIPC) ever performed and will define the role of this novel therapy as a clinical tool. This study will also be the first to define preoperative gene expression profiles associated with poor postoperative outcomes in a control (SHAM) population of children undergoing cardiac surgery. Finally, the role of RIPC in modifying these gene expression profiles will be examined. Therefore, mechanistic insight into the proven ability of RIPC to improve markers of tissue injury, and the expected improvement in clinically relevant endpoints, will be examined.

DETAILED DESCRIPTION:
Remote ischemic preconditioning (RIPC) is a powerful, innate mechanism of protection against ischemia-reperfusion (IR) injury. During the course of previous investigations, it was shown in animal models that transient limb ischemia (our stimulus for generating remote ischemic preconditioning) leads to induction of a portfolio of myocardial genomic responses concerned with stress-response and repair mechanisms, reduces myocardial infarction after prolonged coronary occlusion, protects against cardiopulmonary bypass-induced neural, pulmonary and myocardial damage, and when administered to the recipient, reduces IR injury in the transplanted heart.

In humans, it has been have shown that RIPC downregulates genes responsible for pro-inflammatory pathways concerned with TNFα-signaling, apoptosis and exocytosis in circulating leukocytes, reduces ischemia-induced endothelial dysfunction, and decreases markers of myocardial and lung injury in a pilot study of children undergoing open heart surgery. However, the latter study was not powered to demonstrate differences in anatomic and age-related subgroups, or clinically relevant 'hard' end-points such as ventilation time, intensive care, and length of hospital stay.

Thus, we are now proposing a large-scale clinical study examining genetic predictors of clinically relevant postoperative outcomes, and how they are modified by remote preconditioning.

ELIGIBILITY:
Inclusion Criteria:

* Subject age birth (>36 weeks gestation) to 17 years.
* Underlying cardiac anatomy and planned primary repair with no anticipated residual shunting. Repair must necessitate use of cardiopulmonary bypass.
* Informed consent/assent of subject, parent(s) or legal guardian as appropriate.

Exclusion Criteria:

* Current or recent ischemic insult, defined as vascular occlusion or episode of cardiorespiratory collapse requiring medical intervention occurring within 7 days of enrollment.
* Evidence in any system for organ dysfunction that requires medical intervention.
* Current treatment with systemic anticoagulation therapy or the presence of a bleeding diathesis.
* Presence of important pulmonary or airway disease requiring medical intervention.
* Current or previous (within 10 days of screening) use of systemic corticosteroids.
* Recent (within 7 days of screening) or current documented systemic infection or sepsis.
* Anticipated unavailability of an uninstrumented limb with no anatomic or physiologic abnormality precluding administration of RIPC stimulus using a standard blood pressure cuff.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2008-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Impact of RIPC on length of hospital stay. | Assessed through post-operative hospitalization.

SECONDARY OUTCOMES:
Gene expression patterns associated with effects of RIPC. | Assessed and recorded during the first 24 hours after surgery.
Patterns of baseline gene expression predictive of the clinical and physiologic impact of cardiopulmonary bypass in children (SHAM group only). | Assessed and recorded during the first 24 hours after surgery.
Impact of RIPC on clinical and physiologic markers related to ischemia-reperfusion injury after cardiac surgery in children. | Assessed and recorded serially during the first 48 hours after surgery.
Neurodevelopmental Outcomes (Age < 2 years old at surgery) | Follow-up at 12-18 months post-surgery
  Patients less than a two years of age at the time of surgery will return at 12 -18 months postoperative to be assessed using the BSID- III. During the same visit, parents will complete questionnaires pertaining to their child's behavior and adaptive behavior; the parent version of the Child Behavior Checklist and the parent version of the Vineland Adaptive Behavior Scales - II.
Neurodevelopmental Outcomes (Age 2-6 years old at surgery) | Follow-up at 12-18 months post-surgery
  Patients greater than two years of age at the time of surgery will be assessed using the Wechsler Preschool and Primary Scale of Intelligence-Revised, the Peabody Picture Vocabulary Test - IV and the Beery-Buktenica Developmental Test of Visual-Motor Integration, 5th Edition. Parents will complete questionnaires pertaining to their child's behavior and adaptive behavior; the parent version of the Child Behavior Checklist and the parent version of the Vineland Adaptive Behavior Scales - II.

CONTACTS AND LOCATIONS:
Overall Officials: Brian W. McCrindle, MD MPH, Principal Investigator — The Hospital for Sick Children; Andrew N. Redington, MB, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Brian W. McCrindle, Toronto, Ontario, Canada

REFERENCES:
- [Derived] McCrindle BW, Clarizia NA, Khaikin S, Holtby HM, Manlhiot C, Schwartz SM, Caldarone CA, Coles JG, Van Arsdell GS, Scherer SW, Redington AN. Remote ischemic preconditioning in children undergoing cardiac surgery with cardiopulmonary bypass: a single-center double-blinded randomized trial. J Am Heart Assoc. 2014 Jul 28;3(4):e000964. doi: 10.1161/JAHA.114.000964. PMID 25074698